CLINICAL TRIAL: NCT01254019
Title: A Phase III, Randomized, Double Blind, Placebo-controlled Clinical Study to Assess the Efficacy and Safety of GSK2402968 in Subjects With Duchenne Muscular Dystrophy
Brief Title: A Clinical Study to Assess the Efficacy and Safety of GSK2402968 in Subjects With Duchenne Muscular Dystrophy
Acronym: DMD114044
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114044
Record Dates: First submitted 2010-10-21; First posted 2010-12-06 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2017-09

CONDITIONS: Muscular Dystrophies
Keywords: Duchenne Muscular Dystrophy; DMD; 968; GSK; Duchenne
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GSK2402968 (Experimental): 6mg/kg
  Interventions: Drug: GSK2402968 6mg/kg/week
- Placebo (Experimental): dose-matched
  Interventions: Drug: GSK2402968 6mg/kg/week

INTERVENTIONS:
Drug: GSK2402968 6mg/kg/week — subcutaneous

SUMMARY:
The purpose of this study is to determine whether GSK2402968 is effective in the treatment of ambulant boys with Duchenne muscular dystrophy resulting from a mutation thought to be corrected by exon 51 skipping.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant subjects with Duchenne muscular dystrophy resulting from a mutation/deletion within the DMD gene, confirmed by a state-of-the-art DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation), SCAIP (Single Condition Amplification/Internal Primer) or H-RMCA (High-Resolution Melting Curve Analysis), and correctable by GSK2402968-induced DMD exon 51 skipping.
* Males, aged at least 5 years, and with life expectancy of at least 1 year
* Able to complete 6MWD test with minimal distance of at least 75m at each predrug visit. In addition, results of 6MWD must be within 20% of each other at each pre-drug visit
* Receiving glucocorticoids for a minimum of 6 months immediately prior to screening, with no significant change in total daily dosage or dosing regimen for a minimum of 3 months immediately prior to screening and a reasonable expectation that total daily dosage and dosing regimen will not change significantly for the duration of the study
* QTc <450msec (based on single or average QTc value of triplicate ECGs obtained over a brief recording period), or <480 msec for subjects with Bundle Branch Block. Note: QTc may be either QTcB or QTcF, and machine read or manual overread.
* Subjects, where appropriate, must be willing to use adequate contraception (condoms or abstinence) for the duration of the study and for at least 5 months after the last dose of study drug.
* Willing and able to comply with all protocol requirements and procedures,
* Able to give informed assent and/or consent in writing signed by the subject and/or parent(s)/legal guardian (according to local regulations).
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Any additional missing exon for DMD that cannot be treated with GSK2402968
* Current or history of liver or renal disease or impairment
* Acute illness within 4 weeks of the first anticipated administration of study medication which may interfere with study assessments
* Use of anticoagulants, antithrombotics or antiplatelet agents, previous treatment with investigational drugs, within 6 months of the first administration of study medication; and idebenone or other forms of Coenzyme Q10 within 1 month of the first administration of study medication.
* Current or anticipated participation in any investigational clinical studies
* Positive hepatitis B surface antigen, hepatitis C antibody test (if verified via RIBA or PCA testing), or human immunodeficiency virus (HIV) test at screening,
* Symptomatic cardiomyopathy. If subject has a left ventricular ejection fraction <45% at Screening, the investigator should discuss inclusion of subject in the study with the medical monitor,
* Children in Care. The definition of a Child in Care is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2013-06-28 (Actual); Study Completion 2013-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (45):
- GSK Investigational Site, Buenos Aries, Buenos Aires, Argentina
- GSK Investigational Site, Leuven, Belgium
- Brazil (6):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (2):
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- GSK Investigational Site, Koebenhavn Oe, Denmark
- France (5):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- GSK Investigational Site, Budapest, Hungary
- Italy (4):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Messina, Sicily
- Japan (4):
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Leiden, Netherlands
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Warsaw, Poland
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Esplugues de Llobregat. Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Kaohsiung City, Taiwan
- GSK Investigational Site, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Goemans N, Mercuri E, Belousova E, Komaki H, Dubrovsky A, McDonald CM, Kraus JE, Lourbakos A, Lin Z, Campion G, Wang SX, Campbell C; DEMAND III study group. A randomized placebo-controlled phase 3 trial of an antisense oligonucleotide, drisapersen, in Duchenne muscular dystrophy. Neuromuscul Disord. 2018 Jan;28(1):4-15. doi: 10.1016/j.nmd.2017.10.004. Epub 2017 Dec 6. PMID 29203355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 44 centers in 19 countries from 02 December 2010 to 28 June 2013.
Pre-assignment Details: A total of 186 participants were randomized which included males with a maximum age of 16 years, no adults were included in this study.
Groups:
- Placebo: Participants received single dose of matching placebo sterile solution for subcutaneous injection preferably in the morning over the 48 week treatment period.
- GSK2402968 6mg/kg/Week: Participants received single dose of GSK2402968 6 milligrams per kilogram per week (mg/kg/week) subcutaneous injection preferably in the morning over the 48 week treatment period.
Period: Overall Study
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Started | 61 | 125
Completed | 60 | 121
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- GSK2402968 6mg/kg/Week: Participants received single dose of GSK2402968 6 mg/kg/week subcutaneous injection preferably in the morning over the 48 week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2402968 6mg/kg/Week | Total
Number analyzed (Participants) | 61 | 125 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (2.37) | 8.3 (2.43) | 8.2 (2.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 125 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 1 | 3 | 4
  Asian - East Asian Heritage | 3 | 6 | 9
  Asian - Japanese Heritage | 5 | 9 | 14
  Asian - South East Asian Heritage | 0 | 2 | 2
  White - Arabic/North African Heritage | 4 | 5 | 9
  White - White/Caucasian/European Heritage | 46 | 95 | 141
  White - Mixed Race | 0 | 1 | 1
  Mixed Race | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Muscle Function Using the 6 Minute Walking Distance (6MWD) Test Assessed at Week 48
Description: During the 6MWD, participants were asked to walk, at their own preferred speed, up and down a fixed distance until they were told to stop after 6 minutes. The participants were warned of the time and were told that they may stop earlier if they feel unable to continue. The total distance walked within 6 minutes (or until the participant stopped in case of early termination of the test), the 6MWD, was recorded in meters as well as any falls. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: The Intent-to-Treat (ITT) Population comprised all participants who received at least one dose of study medication and for whom at least one post-Baseline efficacy assessment was available. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 59 | 117
Meters | -52.65 (10.423) | -42.32 (7.378)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.415, Mixed Effect Model for Repeated Measures — Statistical significance was assessed at the 5% level; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = 10.334, 95% CI 2-sided [-14.645 to 35.312]

2. Secondary Outcome: Change From Baseline in the Linearized North Star Ambulatory Assessment (NSAA) Total Score at Week 48
Description: The NSAA is a functional scale devised from the Hammersmith Scale of Motor Ability specifically for use in ambulant children with Duchenne muscular dystrophy (DMD). It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). The scale assesses activities required to remain functionally ambulant (e.g. rise from the floor), activities that can be difficult even early in the disease (e.g. standing on heels) and activities that are known to progressively deteriorate over time (stand from a chair, walk). NSAA total score was achieved by adding the responses of all activities, ranging from 0 to 34, with a score of 34 implying normal function and lower score implying more severe symptoms. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48. A positive change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 58 | 117
Scores on a scale | -6.7 (1.43) | -7.2 (1.01)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.757, Mixed Effect Model for Repeated Measures — Statistical significance (SS) was only to be assessed if a statistically significant difference was observed for the primary and any secondary endpoints higher in the pre-defined hierarchy. Hence conclusions with regards to SS should not be made; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -0.53, 95% CI 2-sided [-3.95 to 2.88]

3. Secondary Outcome: Change From Baseline in the 4 Stair Climb (Ascent) Velocity at Week 48
Description: The participant was asked to ascend four steps. Time was recorded with a stopwatch from the initiation of movement until the participant stood on the fourth step. A flight of steps with handrail was used for this test. Number of stairs ascended per second was calculated as 4 divided by the time to ascend 4 complete stairs. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Stairs per second
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 55 | 111
Stairs per second | -0.12 (0.049) | -0.14 (0.035)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.718, Mixed Effect Model for Repeated Measures — SS was only to be assessed if a statistically significant difference was observed for the primary and any secondary endpoints higher in the pre-defined hierarchy. Hence conclusions with regards to SS should not be made; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -0.021, 95% CI 2-sided [-0.137 to 0.095]

4. Secondary Outcome: Change From Baseline in the 10-meter Walk/Run Velocity at Week 48
Description: The participant was instructed to perform the test bare foot. No aids or orthoses were allowed. The participant was asked to traverse a marked 10-meter measured walkway as quickly as he safely could. Time was recorded to one tenth of a second with a stop watch from when his first foot crossed the start line until when the second foot crossed the finish line. If the wall was touched, it was noted how often. Care was taken to ensure that the participant was safe when completing this test. The assessor walked nearby to provide emergency help if needed, but did not support or provide manual assistance to the participant in any way. If the participant could not complete the 10-meter walk, the total distance was recorded. 10 minute walk/run speed was equal to 10 divided by time taken to complete 10 minute walk/run. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Meters per second
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 58 | 117
Meters per second | -0.20 (0.050) | -0.21 (0.035)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.881, Mixed Effect Model for Repeated Measures — [p-value comment as in outcome 3, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.129 to 0.111]

5. Secondary Outcome: Change From Baseline in the Timed Function Test Rise From Floor at Week 48
Description: The participant stood from a standardized supine position as quickly as possible when told to go. Time was recorded with a stopwatch from the initiation of movement until the assumption of upright standing. No aids or orthoses are allowed. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 44 | 91
Seconds | 7.48 (2.080) | 6.36 (1.463)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.658, Mixed Effect Model for Repeated Measures — No adjustment for multiplicity was made, so p-values should not be used to make conclusions with regards to statistical significance; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -1.115, 95% CI 2-sided [-6.097 to 3.866]

6. Secondary Outcome: Change From Baseline in the 4 Stair Climb (Descent) Velocity at Week 48
Description: The participant was asked to descend four steps. Time was recorded with a stopwatch from the initiation of movement until the participant stood on the fourth step. A flight of steps with handrail was used for this test. Number of stairs descended per second was calculated as 4 divided by the time to descend 4 complete stairs. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Stairs per second
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 55 | 109
Stairs per second | -0.15 (0.052) | -0.11 (0.037)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.513, Mixed Effect Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = 0.041, 95% CI 2-sided [-0.082 to 0.164]

7. Secondary Outcome: Change From Baseline in Muscle Strength (Total Score) at Week 48
Description: Muscle strength was recorded by handheld myometry using a micro force evaluation testing 2 (FET2) myometer. Upper and lower limb proximal muscles were evaluated including knee flexors, knee extensors, elbow flexors, elbow extensors, shoulder abductors and hip flexors. The muscle strength total score (pounds) was the sum of the 12 individual muscle strength tests. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Pounds
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 58 | 118
Pounds | -1.21 (2.729) | -2.18 (1.926)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.769, Mixed Effect Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -0.965, 95% CI 2-sided [-7.446 to 5.516]

8. Secondary Outcome: Kaplan-Meier Estimates for Time to Loss of Ambulation
Description: All participants were ambulant when entered into the study; however they could have become non-ambulant at some time during the study. The date was recorded and the variable time to loss of ambulation was calculated as: time to loss of ambulation = date of loss of ambulation - date of first dose. Median and interquartile range i.e. 1st and 3rd quartile is presented.
Time Frame: Week 48
Population: ITT Population.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Days | NA [NA to NA] — Median, upper limit and lower limit was not reached due to insufficient number of participants with events. | NA [390.0 to NA] — Median and upper limit was not reached due to insufficient number of participants with events.

9. Secondary Outcome: Number of Participants Who Experienced Accidental Falls During 6MWD Assessments at Week 48
Description: The number of accidental falls occurring during the 6MWD were counted. Data has been presented for the number of participants who experienced accidental falls (from 0 to 1) during the 6MWD assessment.
Time Frame: Week 48
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 53 | 103
Participants
  Number of falls=0 | 48 | 102
  Number of falls=1 | 5 | 1

10. Secondary Outcome: Change From Baseline in Creatine Kinase Serum Concentrations at Week 48
Description: Creatine kinase is a muscle-specific enzyme; its level in serum is considered to reflect the extent of muscle damage. In the blood samples drawn to this purpose, the serum level of creatine kinase were measured. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: International units per liter
Groups:
- Placebo: Participants received single dose of matching placebo 1 mL sterile solution for subcutaneous injection preferably in the morning over the 48 week treatment period.
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 60 | 118
International units per liter | -1228.5 (500.59) | -5273.5 (359.05)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo; Test type: Superiority; p = 0.000, Mixed Effect Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = -4044.99, 95% CI 2-sided [-5232.21 to -2857.77]

11. Secondary Outcome: Change From Baseline in Pulmonary Function Test Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1) at Week 48
Description: The FEV1 is the volume of air forcefully exhaled in 1 second, whereas the FVC is the volume of air that can be maximally forcefully exhaled using non-invasive spirometry was conducted to determine actual and percentage values for FVC and FEV1. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Liters
  FVC at Week 48: number analyzed (Participants) | 58 | 121
  FVC at Week 48 | 0.118 (0.1847) | 0.087 (0.2337)
  FEV1 at Week 48: number analyzed (Participants) | 55 | 116
  FEV1 at Week 48 | 0.126 (0.2530) | 0.049 (0.2997)

12. Secondary Outcome: Number of Participants With Identified Mutation: DMD Exon 51 Skip (Upon Muscle Biopsies) at Week 48
Description: Biopsies were taken from their tibialis anterior muscle and few were taken from quadriceps. Total muscle ribonucleic acid (RNA) was isolated from muscle tissue sections and was analyzed by reverse transcriptase polymer chain reaction (RT-PCR). RT-PCR analysis focused on the area flanking the targeted exon 51 was performed to detect specific exon 51 skipping in muscle. Depending on the participants mutation different sets of DMD-gene specific RT and PCR primers were used. Sequence analysis was performed on isolated PCR products to confirm specific exon 51 skip band detection.
Time Frame: Week 48
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 59 | 119
Participants
  DMD Exon 51 skip, Band detected | 48 | 106
  DMD Exon 51 skip, No Band detected | 9 | 9
  DMD Exon 51 skip, No result | 0 | 2
  DMD Exon 51 skip, Not analyzed | 2 | 2

13. Secondary Outcome: Change From Baseline in Pediatric Quality of Life (PedsQL) Total Score at Week 48
Description: PedsQL version 3.0 scale is used to measure pediatric quality of life in children with neuromuscular disorders. The 25-item PedsQL encompasses 3 scales About My/My Childs Neuromuscular Disease (17 items), Communication (3 items), About Our Family Resources (5 items). A 5-point response scale is utilized (where 0=never a problem; 4=almost always a problem). It was assessed both by child and parent. PedsQL total score was calculated by reverse scoring individual items and linearly transforming the score to a 0-100 scale, where higher scores indicated better health-related quality of life. To reverse score individual items, the 0-4 scale items were transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score was then calculated as sum of items divided by number of items answered. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48. A positive change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Scores on a scale
  Assesor child at week 48: number analyzed (Participants) | 57 | 114
  Assesor child at week 48 | 0.52 (11.313) | 1.36 (11.360)
  Assesor parent at week 48: number analyzed (Participants) | 58 | 117
  Assesor parent at week 48 | -0.11 (11.064) | -1.19 (11.269)

14. Secondary Outcome: Change From Baseline in Pulmonary Function Test Peak Cough Flow (PCF) and Peak Flow (PF) at Week 48
Description: The PF also called peak expiratory flow rate (PEFR) is a participants maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a participants ability to breathe out air. PCF was measured for participants wearing a nose clip and performing a maximum cough into a pocket peak flow meter. Baseline was defined as participants randomization assessment at Visit 3 (Day 0). Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Day 0) and Week 48
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Liters per minute
  PF at Week 48: number analyzed (Participants) | 59 | 121
  PF at Week 48 | 25.810 (41.5342) | 11.603 (42.6964)
  PCF at Week 48: number analyzed (Participants) | 59 | 120
  PCF at Week 48 | 22.7 (42.46) | 10.7 (45.04)

15. Secondary Outcome: Number of Participants Who Showed Improvement on Clinician Global Impression of Improvement (CGI-I) Scale at Week 48
Description: The CGI-I is scored based on the clinician's reflection of the participant's current overall clinical condition compared to the overall clinical condition just prior to the initiation of medication use (i.e., the period prior to Randomization). The CGI-I is rated without regard to the clinician's belief that any clinical changes are or are not due to medication and without consideration of the etiology of the symptoms. The CGI-I is measured on a 7-point Likert scale (where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse). The score ranged from 1-7, where lower score indicated more improvement and higher score indicated less improvement.
Time Frame: Week 48
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 57 | 116
Participants
  Very much improved | 0 | 3
  Much improved | 1 | 9
  Minimally improved | 2 | 23
  No change | 27 | 41
  Minimally worse | 20 | 30
  Much worse | 6 | 10
  Very much worse | 1 | 0

16. Secondary Outcome: Change From Baseline in Health Utilities Index (HUI) Scores at Week 48
Description: A 15-item HUI questionnaire assessed Health-related quality of life (HRQoL). Responses from 15-item HUI were used to quantify HRQoL according to 2 health status classification systems, HUI Mark 2 (HUI2) and HUI Mark 3 (HUI3). HUI2 assessed 7 HRQoL dimensions: sensation, mobility, emotion, cognition, self care, pain and fertility. HUI3 assessed 8 HRQoL dimensions: vision, hearing, speech, ambulation, dexterity, emotion, cognition and pain. Both HUI2 (range from -0.03 to 1.0) and HUI3 (range from -0.36 to 1.0) utility scores were calculated using algorithms incorporating community-derived preference weights. A utility value of 1.0 represented perfect health and a utility value of 0.0 represented death. Lowest possible HUI2 score was -0.03 and for HUI3 score was -0.36, where scores less than 0 represented health states considered worse than death. Change from Baseline was calculated by subtracting Baseline value from Week 48 value. A positive change from Baseline indicated improvement.
Time Frame: Baseline (Randomization Visit, Day 0) and Week 48
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Scores on a scale
  HUI2 at Week 48: number analyzed (Participants) | 53 | 112
  HUI2 at Week 48 | -0.052 (0.0190) | -0.023 (0.0133)
  HUI3 at Week 48: number analyzed (Participants) | 56 | 116
  HUI3 at Week 48 | -0.061 (0.0266) | -0.056 (0.0188)
Statistical Analysis 1: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo, HUI2 at Week 48; Test type: Superiority; p = 0.207, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = 0.0288, 95% CI 2-sided [-0.0161 to 0.0738]
Statistical Analysis 2: Comparison: Placebo vs GSK2402968 6mg/kg/Week; GSK2402968 6mg/kg/week Vs Placebo, HUI3 at Week 48; Test type: Superiority; p = 0.880, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; Model included terms for treatment, visit, treatment by visit, country grouping, Baseline and Baseline by visit; Mean Difference (Net) = 0.0048, 95% CI 2-sided [-0.0580 to 0.0676]

17. Secondary Outcome: Number of Participants With Adverse Events (AE) and Severe Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect.
Time Frame: Up to Follow-up (Week 68)
Population: The Safety Population comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  Any AE | 58 | 123
  Any SAE | 5 | 13

18. Secondary Outcome: Number of Participants With Vital Sign Data for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) and Heart Rate (HR) of Potential Clinical Concern (PCC) at Any Visit Post-Baseline
Description: Blood pressure SBP, DBP and HR were recorded after five minutes of rest in a semi-supine position. The following changes from Baseline (Day 0) in vital signs were considered to be of potential clinical concern: DBP was defined as high (increase from Baseline >=20 and >=40 millimeters of mercury [mmHg] and low (decrease from Baseline >=20 and >=40 mmHg), SBP high (increase from Baseline >=10 and >=20 mmHg and low (decrease from Baseline >=10 and >=20 mmHg) and for HR high (increase from Baseline >=20 and >=40 beats per minute [bpm] and low (decrease from Baseline >=20 and >=40 bpm). Only those parameters for which a value of PCC was reported at any visit post-Baseline is presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  DBP, High at any visit post-Baseline | 22 | 52
  HR, low at any visit post-Baseline | 19 | 49
  HR, high at any visit post-Baseline | 18 | 32
  SBP, low at any visit post-Baseline | 8 | 7
  SBP, high at any visit post-Baseline | 28 | 72

19. Secondary Outcome: Number of Participants With Abnormal-clinically Significant Electrocardiogram (ECG) Findings at Any Visit Post-Baseline
Description: ECG measurements were carried out and the clinical interpretation of the ECG by the investigator was recorded as normal, abnormal but not clinically significant and abnormal clinically significant. The PCC ranges include, QT interval corrected for heart rate by Bazett's formula (QTcB) or QT interval corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds and any increase from Baseline of QTcB or QTcF. Participants were categorized as abnormal clinically significant based on the investigator's judgment and PCC ranges. Data has been presented for number of participants with abnormal clinically significant findings at any visit post-Baseline.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants | 0 | 5

20. Secondary Outcome: Number of Participants With Hematology Parameters of PCC at Any Visit Post-Baseline
Description: Laboratory samples were collected for analysis of hematology parameters. The PCC values for hematology parameters: hematocrit was 1.02 x Upper limit of normal (ULN), for hemoglobin was 1.03 x ULN, for lymphocytes was 0.81 x lower limit of normal (LLN), for platelet count was 0.67 x LLN and 1.57 x ULN, for total neutrophils was 0.83 x LLN, and that for white blood cell count was 0.67 x LLN and value of 1.82 x ULN. Only those parameters for which a value of PCC was reported at any visit post-Baseline have been presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  Hematocrit > reference range high | 12 | 27
  Hemoglobin > reference range high | 2 | 6
  Lymphocytes < reference range low | 6 | 9
  Platelet count > reference range high | 1 | 0
  Platelet count < reference range low | 0 | 1
  Total neutrophils < reference range low | 8 | 9
  White blood cell count < reference range low | 3 | 4

21. Secondary Outcome: Number of Participants With Coagulation Parameters of PCC at Any Visit Post-Baseline
Description: Laboratory samples were collected for analysis of coagulation parameters. The PCC values for coagulation parameters activated partial thromboplastin time (aPTT) was 1.5 x ULN and aPTT ratio also known as international normalized ration (INR) was 1.2 x ULN. Only those parameters for which a value of PCC was reported at any visit post-Baseline is presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  aPTT > reference range high | 6 | 6
  INR > reference range high | 11 | 32

22. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of PCC at Any Visit Post-Baseline
Description: Laboratory samples were collected for analysis of chemistry parameters. The PCC values for chemistry parameters for alanine amino transferase (ALT) plus total bilirubin (TB) was >=1.5 x ULN for TB and >=2 x ULN for ALT, for albumin was 0.86 x LLN, for asparatate amino transferase (AST) was >=2 x ULN, for calcium was 0.91 x LLN and 1.06 x ULN, for glucose was 0.71 x LLN and 1.41 x ULN, for phosphorus was 0.80 x LLN and 1.14 x ULN, for sodium was 0.96 x LLN and 1.03 x ULN, for potassium was 0.86 x LLN and 1.10 x ULN and that for alkaline phosphatase was >=2x ULN. Only those parameters for which a value of PCC was reported at any visit post-Baseline is presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  ALT plus TB > reference range high | 0 | 2
  ALT > reference range high | 61 | 125
  Albumin < reference range low | 0 | 1
  AST > reference range high | 61 | 125
  Calcium > reference range high | 1 | 3
  Calcium < reference range low | 0 | 3
  Glucose > reference range high | 3 | 5
  Glucose < reference range low | 0 | 2
  Phosphorus > reference range high | 1 | 8
  Sodium > reference range high | 2 | 9
  Potassium > reference range high | 0 | 0
  Potassium < reference range low | 0 | 0
  Alkaline phosphatase > reference range high | 0 | 0

23. Secondary Outcome: Number of Participants With Urinalysis Data Outside the Reference Range (>Reference Range High) at Any Visit Post- Baseline
Description: Urine samples were collected for analysis of abnormal urine parameters. Quantitative examination included the assessment for urine albumin excretion rate, urine alpha-1-microglobulin, urine creatinine excretion-24 hour and urine protein excretion-24 hour. Only those parameters for which a value of >reference range high was reported at any visit post-Baseline is presented.
Time Frame: Up to Week 48
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 61 | 125
Participants
  Urine Albumin excretion rate > reference range: number analyzed (Participants) | 12 | 93
  Urine Albumin excretion rate > reference range | 1 | 15
  Urine Protein excretion -24 hour > reference range: number analyzed (Participants) | 12 | 96
  Urine Protein excretion -24 hour > reference range | 4 | 54

24. Secondary Outcome: Plasma Concentrations of GSK2402968 Following Subcutaneous Administration
Description: Blood samples for pharmacokinetic assessment were taken at Week 0 (Randomization) at 0.5, 1, 3 hours post-dose and at Week 8,12, 24, 36 and 47 at pre-dose, and between 1 and 4 hours post-dose. Data has been presented for plasma concentrations of GSK2402968 following subcutaneous administration.
Time Frame: Randomization (Week 0 at 0.5, 1 and 3 hours), Week 8 (pre-dose, 1-4 hours), Week 12 (pre-dose, 1-4 hours), Week 24 (pre-dose, 1-4 hours), Week 36 (pre-dose, 1-4 hours), Week 47 (pre-dose, 1-4 hours)
Population: The Pharmacokinetic Population comprised all participants who were randomized to the study and from whom at least one blood sample was obtained for assessment of GSK2402968 concentration. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Nanograms per millimeter
Arm/Group | GSK2402968 6mg/kg/Week
Number analyzed (Participants) | 125
Nanograms per millimeter
  Week 0, 0.5 hours: number analyzed (Participants) | 120
  Week 0, 0.5 hours | 3349.595 [572.07 to 10408.94]
  Week 0, 1 hour: number analyzed (Participants) | 122
  Week 0, 1 hour | 4946.950 [1094.90 to 13159.51]
  Week 0, 3 hour: number analyzed (Participants) | 121
  Week 0, 3 hour | 5932.740 [1794.00 to 12765.26]
  Week 8, Pre-dose: number analyzed (Participants) | 47
  Week 8, Pre-dose | 12.730 [0.00 to 4424.28]
  Week 8, 1-4 hours: number analyzed (Participants) | 47
  Week 8, 1-4 hours | 5100.220 [7.62 to 10471.64]
  Week 12, Pre-dose: number analyzed (Participants) | 47
  Week 12, Pre-dose | 19.090 [4.60 to 50.95]
  Week 12, 1-4 hours: number analyzed (Participants) | 47
  Week 12, 1-4 hours | 5613.040 [10.89 to 10583.33]
  Week 24, Pre-dose: number analyzed (Participants) | 49
  Week 24, Pre-dose | 40.920 [0.00 to 186.87]
  Week 24, 1-4 hours: number analyzed (Participants) | 49
  Week 24, 1-4 hours | 6141.580 [40.65 to 11902.15]
  Week 36, Pre-dose: number analyzed (Participants) | 38
  Week 36, Pre-dose | 55.185 [22.64 to 6590.81]
  Week 36, 1-4 hours: number analyzed (Participants) | 37
  Week 36, 1-4 hours | 5755.950 [68.84 to 12967.56]
  Week 47, Pre-dose: number analyzed (Participants) | 106
  Week 47, Pre-dose | 61.395 [3.86 to 5922.31]
  Week 47, 1-4 hours: number analyzed (Participants) | 99
  Week 47, 1-4 hours | 5266.240 [46.42 to 13841.11]

ADVERSE EVENTS:
Time Frame: Up to Follow-up (Week 68).
Description: The Safety Population was used for analysis.
Arm/Group | Placebo | GSK2402968 6mg/kg/Week
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/125
Serious Adverse Events (participants affected / at risk) | 5/61 | 13/125
Other Adverse Events (participants affected / at risk) | 54/61 | 119/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | GSK2402968 6mg/kg/Week (N=125)
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1
Cardiac fibrillation (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Spinal pain (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | GSK2402968 6mg/kg/Week (N=125)
Injection site erythema (General disorders) | 4 | 62
Injection site discolouration (General disorders) | 2 | 41
Pyrexia (General disorders) | 15 | 27
Injection site pain (General disorders) | 2 | 23
Injection site reaction (General disorders) | 1 | 24
Injection site bruising (General disorders) | 6 | 11
Injection site induration (General disorders) | 0 | 17
Injection site pruritus (General disorders) | 0 | 17
Injection site haematoma (General disorders) | 2 | 9
Injection site atrophy (General disorders) | 0 | 9
Injection site urticaria (General disorders) | 0 | 9
Injection site swelling (General disorders) | 0 | 8
Nasopharyngitis (Infections and infestations) | 25 | 38
Upper respiratory tract infection (Infections and infestations) | 8 | 15
Gastroenteritis (Infections and infestations) | 5 | 15
Rhinitis (Infections and infestations) | 3 | 10
Influenza (Infections and infestations) | 4 | 7
Ear infection (Infections and infestations) | 5 | 4
Pharyngitis (Infections and infestations) | 4 | 5
Bronchitis (Infections and infestations) | 4 | 4
Vomiting (Gastrointestinal disorders) | 13 | 28
Diarrhoea (Gastrointestinal disorders) | 9 | 23
Abdominal pain (Gastrointestinal disorders) | 7 | 14
Abdominal pain upper (Gastrointestinal disorders) | 3 | 9
Proteinuria (Renal and urinary disorders) | 11 | 42
Haematuria (Renal and urinary disorders) | 5 | 21
Fall (Injury, poisoning and procedural complications) | 12 | 26
Contusion (Injury, poisoning and procedural complications) | 7 | 8
Excoriation (Injury, poisoning and procedural complications) | 3 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 7
Protein urine present (Investigations) | 4 | 17
Red blood cells urine positive (Investigations) | 4 | 14
Cystatin C increased (Investigations) | 2 | 14
Red blood cells urine (Investigations) | 4 | 11
Urine protein/creatinine ratio increased (Investigations) | 2 | 11
Blood fibrinogen decreased (Investigations) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 10
Headache (Nervous system disorders) | 11 | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7
Ear pain (Ear and labyrinth disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.